CLINICAL TRIAL: NCT01044017
Title: A Single-center, Double-blind, Randomized, Cross-over, Placebo-controlled, Single-dose Study to Investigate Glycemic Parameters of Efficacy During 24 Hours, Safety/ Tolerability and Pharmacokinetics of Two Dose Levels of RO4998452 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Single Doses of RO4998452 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: BP22764; 2009-013124-23
Record Dates: First submitted 2009-11-17; First posted 2010-01-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A (Experimental)
  Interventions: Drug: RO4998452
- B (Experimental)
  Interventions: Drug: RO4998452
- C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — single oral dose
  Arms: C
Drug: RO4998452 — single oral doses
  Arms: A; B

SUMMARY:
This randomized, double-blind, placebo-controlled, cross-over study will evaluate the glucose concentration and other glycemic parameters of efficacy, and the safety and tolerability and pharmacokinetics of single oral doses of RO4998452 in patients with diabetes mellitus type 2. On 3 treatment days a week apart, patients will each receive orally one of 2 dose levels of RO4998452 or placebo. Anticipated time of study treatment is 3 weeks. Target sample size is <50.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-75 years of age
* Type 2 diabetes mellitus, diagnosed for at least 3 months at screening
* Treatment with diet and exercise
* BMI between 27 and 40 kg/m2

Exclusion Criteria:

* Type 1 diabetes
* History of ketoacidosis, hyperosmolar coma, or lactic acidosis
* Renal disease or renal dysfunction
* Evidence of significant diabetic complication
* Currently or within 3 months prior to screening treated with any oral or injectable anti-diabetic agents (exception: insulin injection in emergency situation)
* History of anti-diabetic triple therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Effect on postprandial plasma glucose concentration | Following meal 13 hours after dosing

SECONDARY OUTCOMES:
Mean postprandial daily plasma glucose concentration (3 consecutive meals) | 25 hours
Mean daily blood glucose concentration, pre-meal plasma glucose concentration, plasma insulin concentration | Assessments up to 25 hours after dosing
Urinary glucose excretion | Assessments up to 25 hours after dosing
Safety and tolerability: AEs, laboratory parameters | AEs throughout study, laboratory assessments on 3 treatment days and on follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Strasbourg, France